CLINICAL TRIAL: NCT04587830
Title: Phase 1-2 Trial of ADI-PEG 20 Plus Radiotherapy and Temozolomide in Subjects With Newly Diagnosed Glioblastoma Multiforme (GBM)
Brief Title: ADI-PEG 20 Plus Radiotherapy and Temozolomide in Subjects With Glioblastoma Multiforme
Acronym: GBM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POLARIS2020-001
Record Dates: First submitted 2020-09-04; First posted 2020-10-14 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma Multiforme (GBM)
Keywords: argininosuccinate synthetase; arginine; arginine deiminase
MeSH Terms: conditions — Glioblastoma | interventions — ADI PEG20; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADI-PEG 20 plus Radiotherapy and Temozolomide (Experimental): ADI-PEG 20 Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM)
  Radiotherapy Dose: 60 Gy in 30 daily (Monday-Friday) fractions of 2 Gy each; to start within 4 weeks of surgery (diagnostic and/or resection)
  Temozolomide Dose: 75 mg/m2 daily during radiotherapy; 150-200 mg/m2 for 5 days every 4 weeks (1 cycle) x 6 cycles during maintenance period Route of Administration: oral or intravenous
  Interventions: Drug: ADI-PEG 20; Drug: Temozolomide
- Placebo plus Radiotherapy and Temozolomide (Placebo Comparator): Placebo Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM)
  Radiotherapy Dose: 60 Gy in 30 daily (Monday-Friday) fractions of 2 Gy each; to start within 4 weeks of surgery (diagnostic and/or resection)
  Temozolomide Dose: 75 mg/m2 daily during radiotherapy; 150-200 mg/m2 for 5 days every 4 weeks (1 cycle) x 6 cycles during maintenance period Route of Administration: oral or intravenous
  Interventions: Drug: Temozolomide; Drug: Placebo

INTERVENTIONS:
Drug: ADI-PEG 20 — Investigational Medicine
  Arms: ADI-PEG 20 plus Radiotherapy and Temozolomide
Drug: Temozolomide — Radiotherapy and TMZ are standard front-line therapy for newly diagnosed GBM.
Drug: Placebo — Investigational Medicine
  Arms: Placebo plus Radiotherapy and Temozolomide

SUMMARY:
A randomized, double-blind, placebo-controlled study. Weekly ADI-PEG 20 (36 mg/m2) or placebo will be combined with Stupp Protocol (Stupp 2005) radiotherapy and TMZ

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study. Weekly ADI-PEG 20 (36 mg/m2) or placebo will be combined with Stupp Protocol (Stupp 2005) radiotherapy and TMZ as noted for the Phase 1 portion. Furthermore, ADI-PEG 20 or placebo treatment may continue after adjuvant TMZ if there is no progressive disease, for up to a total of 2 years of ADI-PEG 20 or placebo treatment. In addition, after 24 weeks (6 cycles) subjects may also continue adjuvant TMZ along with ADI-PEG 20 or placebo, in the absence of disease progression, as noted above, if clinically indicated in the investigator's judgement. MRI is to be performed post-surgery(biopsy), and then at 1, 3 and 6 months after completion of radiotherapy and then every 3 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, histologically confirmed glioblastoma, IDH-wildtype and the WHO Grade 4 of astrocytoma, IDH-mutant by WHO 2021 classification of brain tumors, non-resectable or partially resected or resected.
2. Age 20 - 75 years.
3. Karnofsky Performance Status (KPS) ≥ 60.
4. Expected life expectancy ≥16 weeks.
5. Stable or decreasing corticosteroids (5 mg/day dexamethasone or equivalent) within 5 days before the first dose of ADI-PEG 20.
6. No prior systemic therapy, immunotherapy, investigational agent, or radiation therapy.
7. Recovered from any prior surgery and no major surgery within 2 weeks of initiating treatment (other than GBM surgery). Surgery for placement of vascular access devices is acceptable.
8. Female subjects and male subjects must be asked to use appropriate contraception for both the male and female for the duration of the study and for at least 30 days after the last administration of ADI-PEG 20 or placebo and at least 6 months after the last administration of TMZ. Male partners of female subjects and female partners of male subjects must agree to use two forms of contraception or agree to refrain from intercourse for the duration of the study if they are of childbearing potential. Females of childbearing potential must not be pregnant at the start of the study, and a serum human chorionic gonadotropin (HCG) pregnancy test must be negative before entry into the study. If positive HCG pregnancy test, further evaluation to rule out pregnancy must be performed according to GCP before this subject is deemed eligible. Females not of childbearing potential must be post-menopausal (defined as cessation of regular menstrual period for at least 12 months).
9. Informed consent must be obtained prior to study initiation.
10. No concurrent investigational studies are allowed.
11. Absolute neutrophil count (ANC) ≥ 1500/μL.
12. Platelets ≥ 100,000/μL.
13. Serum uric acid ≤ 8 mg/dL (with or without medication control).
14. Creatinine clearance must be ≥ 40 mL/min/1.73 m2 (calculated using the Cockcroft-Gault equation: calculated creatinine clearance = (140-age (yrs)) × body weight (kg) (×0.85 if female) / 72 × serum creatinine (mg/dl).
15. Total bilirubin ≤ 2 x upper limit of normal.
16. ALT and AST ≤ 3 x upper limit of normal, unless liver metastases present then ≤ 5 x upper limit normal.

Exclusion Criteria:

1. Serious infection requiring treatment with systemically administered antibiotics at the time of study entrance, or an infection requiring systemic antibiotic therapy within 7 days prior to the first dose of study treatment.
2. Pregnancy or lactation.
3. Expected non-compliance.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, or psychiatric illness, social situations that would limit compliance with study requirements.
5. Subjects with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present or in the opinion of the investigator will not affect patient outcome.
6. Subjects who had been treated with ADI-PEG 20 previously.
7. History of uncontrolled seizure disorder not related to underlying cancer.
8. Known HIV positivity, or active hepatitis B infection, or active hepatitis C infection (testing not required).
9. Allergy to pegylated compounds.
10. Allergy to E. coli drug products (such as GMCSF).
11. Allergy to TMZ or any of its components.
12. History of hypersensitivity to dacarbazine.
13. Placement of Gliadel wafer at surgery.
14. Having a co-existing condition requiring systemic treatment with either corticosteroids or immunosuppressive medication.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Through study completion, 2.5 year anticipated
  In the ADI-PEG 20 treated arm compared to the placebo arm, and determine if predefined patient subtypes or associated biomarkers uniquely benefit from the treatment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Through study completion, 2.5 year anticipated
  PFS will be reported as the time subject experience from the start of treatment to disease progression or death, measured in month.
Duration of response (DOR) | Through study completion, 2.5 year anticipated
  DOR is reported as the time from when the tumor begins to respond to treatment (first occurrence of CR or PR) until disease progression or deterioration occurs (diagnosis of disease progression), measured in month.
Tumor response rate | Through study completion, 2.5 year anticipated
  Response rate is usually measured in percentage (%). It represents the proportion of subjects whose tumors achieve partial or complete response among those who received treatment.
Safety and tolerability of ADI-PEG 20 | Through study completion, 2.5 year anticipated
  Safety and tolerability in the ADI-PEG 20 treated arm compared to the placebo arm.
  Incidence of Treatment-Emergent Adverse Events from first dose to time of progression or death.
  The severity of all AEs will be assessed according to the NCI CTCAE Scale version 5.
Pharmacokinetics of ADI-PEG 20 | Up to week 52 or End of treatment visit
  ADI-PEG 20 Plasma Concentrations are measured over time, samples are collected before the dosing, and on week 0, 1, 2, 4, 6, 8, 10, 12, 16, 20, 24, 28 and 32, then every 4 weeks until week 52 or End of treatment visit.
Pharmacodynamics of ADI-PEG 20 | Up to week 52 or End of treatment visit
  Citrulline and Arginine plasma concentrations are measured over time, samples are collected before the dosing, and on week 0, 1, 2, 4, 6, 8, 10, 12, 16, 20, 24, 28 and 32, then every 4 weeks until week 52 or End of treatment visit.
Immunogenicity of ADI-PEG 20 | Up to week 52 or End of treatment visit
  Antibodies for ADI-PEG 20, Anti-PEG antibodies are measured in plasma over time, samples are collected before the dosing, and on week 0, 1, 2, 4, 6, 8, 10, 12, 13, 16, 20, 24, then once a month for three months, followed by once every three months until week 52 or End of treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chen Wei, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (10):
- South Korea (5):
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul, Seocho-gu
  - Severance Hospital Yonsei University, Seoul, Seodaemun-gu
  - Seoul National University Bundang Hospital, Gyeonggi-do, Seongnam
- Taiwan (5):
  - Chang Gung-Medical Foundation-Keelung (CGMF-KL), Keelung, Anle Dist
  - Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District, Guishan Dist
  - Chang Gung Medical Foundation-Kaohsiung, Kaohsiung City, Niaosong Dist
  - Mackay Memorial Hospital-Tamsui Branch, New Taipei City, Tamsui Dist
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist

IPD SHARING:
Plan to Share IPD: No